CLINICAL TRIAL: NCT06296641
Title: Leveraging COmmunity Partnered nEeds Navigation to Reduce Unmet Health-related Social Needs Among Caregivers for Adolescent and Younger Adult Cancer Survivors
Brief Title: Needs Navigation for Caregivers of AYAs
Acronym: Cope-CAYAC
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: funding pause
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Melissa Beauchemin, Assistant Professor of Nursing, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAU9477
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cancer in Adolescence
Keywords: Cancer; Adolescents; Young adults; Financial needs; Social needs; Minority health; Caregivers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants who screen positive all move forward to receive the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Needs Navigation Intervention (Experimental): Individuals who screen positive will all move forward to receive this intervention. This includes connection to community partners with financial education and easily accessible resources, and a vocational navigation and support consultation for caregivers for 6-months.
  Interventions: Behavioral: Needs navigation intervention

INTERVENTIONS:
Behavioral: Needs navigation intervention — The investigator anticipates that this will include a baseline financial, education and vocational assessment, likely using a virtual platform. Participants who screen positive will be connected to community resources and for consultation. There will be a 1-month, 3-month and 6-month check-in to address any financial concerns through additional counseling/navigation.

SUMMARY:
The overall aim of the study is to address unmet health-related social needs and reduce outcome disparities among AYA (adolescent and young adult) cancer survivors. Aim 1 aimed to refine a needs navigation model in partnership with expert consultants. Aim 2 and 3 will involve the deployment and pilot testing of the adapted needs navigation intervention among caregivers of younger AYAs with cancer.

DETAILED DESCRIPTION:
Financial toxicity, the negative personal financial impact of healthcare, is a highly prevalent adverse effect of cancer treatment, and AYA cancer survivors experience disproportionately higher rates of financial toxicity compared to older cancer survivors. Financial toxicity is associated with poorer overall survival and bankruptcy, and AYA survivors are 10 times more likely to file for bankruptcy than older cancer survivors. Thus, financial toxicity and unmet HRSN (health-related social needs) are key contributors to employment and health outcome disparities seen among AYA survivors living in areas of persistent poverty.

The study team has focused on addressing unmet HRSN and reducing outcome disparities among AYA cancer survivors, many of whom live in areas of persistent poverty. The investigators have adapted a model of financial navigation that reduces financial toxicity among older adults with cancer, informed by qualitative research among Spanish- and English-speaking AYAs and their caregivers from the local community. The investigators have identified community and clinical partners poised to address these unique unmet needs. These partners have expertise in educational navigation and caregiver community resources - both cited as unmet needs in our pilot study. Using mixed methods, this study will refine (Aim 1 - already completed) and pilot test (Aims 2 and 3) a tailored version of the intervention among 30 English and Spanish-speaking caregivers of younger AYAs who screen positive for severe financial toxicity or unmet HRSN.

ELIGIBILITY:
Inclusion Criteria: We are enrolling dyads (AYA and caregivers) for this study.

AYA patient participants:

* Age 15 - 26 years old
* English or Spanish-speaking
* In between 3-months of diagnosis of cancer date and up to 1-year post-treatment completion without progression or recurrence of cancer

Caregiver/financial partner participants:

* Parent or financially-responsible adult of non-adult AYA (<18 years) OR
* Identified by the AYA as caregiver, parent, or partner who is financially-responsible or a financial partner for AYA

Exclusion Criteria:

* Dyad with caregiver or younger AYA that previously participated in study AAAU2405
* Unable to complete financial survey questions or contraindicated (as outlined in Protection of Human Subjects)
* Dyad with younger AYAs who are enrolled on hospice or receiving other end-of-life care

Ages: 15 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of (OR percentage of) participants who completed the intervention | up to 6 months
  This is to assess the feasibility of intervention completion. Intervention completion is defined as participants who have demonstrated contact for consultation and with community partners at any time before the end of 6 months.
Percentage of eligible participants who consented to be in study | Up to 6 months
  This is to measure interest and the need for help by the intervention that can provide caregiver / patient financial education and navigation

SECONDARY OUTCOMES:
Personal Financial Wellness Scale (PFWS) / Comprehensive Score of Financial Toxicity (COST measure) | Baseline, 6-months
  The PFWS/ COST is a participant-reported outcome measure that describes financial distress in cancer patients or their caregivers.

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zafar SY, Peppercorn JM, Schrag D, Taylor DH, Goetzinger AM, Zhong X, Abernethy AP. The financial toxicity of cancer treatment: a pilot study assessing out-of-pocket expenses and the insured cancer patient's experience. Oncologist. 2013;18(4):381-90. doi: 10.1634/theoncologist.2012-0279. Epub 2013 Feb 26. PMID 23442307
- [Background] Altice CK, Banegas MP, Tucker-Seeley RD, Yabroff KR. Financial Hardships Experienced by Cancer Survivors: A Systematic Review. J Natl Cancer Inst. 2016 Oct 20;109(2):djw205. doi: 10.1093/jnci/djw205. Print 2017 Feb. PMID 27754926
- [Background] Yabroff KR, Dowling EC, Guy GP Jr, Banegas MP, Davidoff A, Han X, Virgo KS, McNeel TS, Chawla N, Blanch-Hartigan D, Kent EE, Li C, Rodriguez JL, de Moor JS, Zheng Z, Jemal A, Ekwueme DU. Financial Hardship Associated With Cancer in the United States: Findings From a Population-Based Sample of Adult Cancer Survivors. J Clin Oncol. 2016 Jan 20;34(3):259-67. doi: 10.1200/JCO.2015.62.0468. Epub 2015 Dec 7. PMID 26644532
- [Background] Ramsey SD, Bansal A, Fedorenko CR, Blough DK, Overstreet KA, Shankaran V, Newcomb P. Financial Insolvency as a Risk Factor for Early Mortality Among Patients With Cancer. J Clin Oncol. 2016 Mar 20;34(9):980-6. doi: 10.1200/JCO.2015.64.6620. Epub 2016 Jan 25. PMID 26811521
- [Background] Parsons SK, Keegan THM, Kirchhoff AC, Parsons HM, Yabroff KR, Davies SJ. Cost of Cancer in Adolescents and Young Adults in the United States: Results of the 2021 Report by Deloitte Access Economics, Commissioned by Teen Cancer America. J Clin Oncol. 2023 Jun 10;41(17):3260-3268. doi: 10.1200/JCO.22.01985. Epub 2023 Feb 24. PMID 36827624
- [Background] Danhauer SC, Canzona M, Tucker-Seeley RD, Reeve BB, Nightingale CL, Howard DS, Puccinelli-Ortega N, Little-Greene D, Salsman JM. Stakeholder-informed conceptual framework for financial burden among adolescents and young adults with cancer. Psychooncology. 2022 Apr;31(4):597-605. doi: 10.1002/pon.5843. Epub 2021 Nov 5. PMID 34699110
- [Background] Guy GP Jr, Yabroff KR, Ekwueme DU, Smith AW, Dowling EC, Rechis R, Nutt S, Richardson LC. Estimating the health and economic burden of cancer among those diagnosed as adolescents and young adults. Health Aff (Millwood). 2014 Jun;33(6):1024-31. doi: 10.1377/hlthaff.2013.1425. PMID 24889952
- [Background] Shah K, Zafar SY, Chino F. Role of financial toxicity in perpetuating health disparities. Trends Cancer. 2022 Apr;8(4):266-268. doi: 10.1016/j.trecan.2021.12.007. Epub 2022 Jan 13. PMID 35034866
- [Background] Beauchemin MP, Solomon S, Michaels CL, McHenry K, Turi E, Khurana R, Sanabria G. Toward identification and intervention to address financial toxicity and unmet health-related social needs among adolescents and emerging adults with cancer and their caregivers: A cross-cultural perspective. Cancer Med. 2024 Apr;13(8):e7197. doi: 10.1002/cam4.7197. PMID 38659403
- [Background] Beauchemin MP, DeStephano D, Raghunathan R, Harden E, Accordino M, Hillyer GC, Kahn JM, May BL, Mei B, Rosenblat T, Law C, Elkin EB, Kukafka R, Wright JD, Hershman DL. Implementation of Systematic Financial Screening in an Outpatient Breast Oncology Setting. JCO Clin Cancer Inform. 2023 Mar;7:e2200172. doi: 10.1200/CCI.22.00172. PMID 36944141